CLINICAL TRIAL: NCT05655910
Title: Enhanced Nutritional Optimization in LVAD (ENOL) Trial
Brief Title: Enhanced Nutritional Optimization in LVAD Trial
Acronym: ENOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAT9591
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure; Gut Microbiome; Nutritional Deficiency
Keywords: Left Ventricular Assist Device (LVAD); Advanced Heart Failure; Mechanical Circulatory Support; Infection; Gut Microbiome
MeSH Terms: conditions — Heart Failure; Malnutrition; Infections

STUDY DESIGN:
Intervention Model Description: Three parallel comparison groups will be created based on assessment of nutritional status and randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Not malnourished) - 3 products per day (Experimental): Patients assessed as well-nourished based on AND-ASPEN criteria and randomized to receive 3 Ensure Surgery Immunonutrition shake per day during the days from consent to LVAD implantation.
  Interventions: Dietary Supplement: Ensure Surgery Immunonutrition shake
- Group 1 (Not malnourished) - 1 product per day (Experimental): Patients assessed as well-nourished based on AND-ASPEN criteria and randomized to receive 1 Ensure Surgery Immunonutrition shake per day during the days from consent to LVAD implantation.
  Interventions: Dietary Supplement: Ensure Surgery Immunonutrition shake
- Group 2 (at risk/malnourished) (Experimental): Patients assessed as at risk for malnourishment or malnourished based on AND-ASPEN criteria automatically assigned to receive 3 Ensure Surgery Immunonutrition shake per day during the days from consent to LVAD implantation.
  Interventions: Dietary Supplement: Ensure Surgery Immunonutrition shake

INTERVENTIONS:
Dietary Supplement: Ensure Surgery Immunonutrition shake — Nutrition shake to support immune health and recovery from surgery.

SUMMARY:
The goal of this clinical trial is to assess whether a peri-operative intervention with nutritional immune modulating intervention (Ensure Surgery Immunonutrition shake) has beneficial effects on the complex interplay between gut microbiome, systemic inflammation and malnutrition that is commonly present in advanced heart failure and the adverse events associated with left ventricular assist device (LVAD) placement in hospitalized advanced heart failure patients awaiting LVAD implantation. The main questions it aims to answer are:

* Will pre-surgical supplementation with Ensure Surgery affect gut microbial composition and levels of inflammation among heart failure patients undergoing LVAD implantation?
* Will pre-surgical supplementation with Ensure Surgery affect post-surgical morbidity (e.g., infections, intensive care unit length of stay (LOS)) and mortality? Participants will be evaluated for malnutrition and will be given Ensure Surgery Immunonutrition shake to drink in the days preceding their LVAD surgery. Blood and stool samples will be collected at prespecified timepoints before and after surgery.

Researchers will compare malnourished participants drinking Ensure Surgery 3/day with well-nourished participants randomized to drink either 1/day or 3/day to see if any of the above supplementation strategies change the gut microbial composition, levels of inflammation, and post-surgical morbidity and mortality.

DETAILED DESCRIPTION:
Heart failure (HF) has an estimated prevalence of >37.7 million individuals globally. In the US alone, which is projected to increase by 46% between the years 2012 and 2030. Despite significant advances in HF medical and device therapies, patient prognosis after their first HF hospital admission is poor, with a <50% survival rate at five years and significant proportion of patients progressing from chronic stable disease to advanced HF state. Once advanced HF ensues, LVADs are one of the two main treatment modalities that can meaningfully improve survival in this patient population.

Chronic systemic inflammation is commonly observed in HF and is believed to be directly related to its pathogenesis. Recently, perturbations in the gut microbiota known as "gut dysbiosis" and impairment of gut mucosal barriers, facilitating entry of endotoxins and gut metabolites into the circulation, have also been observed in HF patients. Elevated levels of circulating endotoxins and bacterial bi-products enhance systemic inflammation, thereby contributing to progression of HF to more advanced disease state. Gut microbial perturbations may also alter enterocyte structure and function resulting in gastrointestinal dysmotility, nutrient malabsorption and eventually malnutrition.

Malnutrition is frequent in HF (as high as 62%), is associated with higher rates of mortality, hospital readmissions and an increased risk of adverse early postoperative outcomes. Infections are the most common complications following LVAD, affecting >50% of HF patients, contributing significantly to postoperative mortality, increased length-of stay (LOS) and hospital readmissions. The pre-operative period may represent an attractive time window in which to optimize HF patients, correct deficiencies, and enhance immune defense mechanisms before surgery. This period allows to act upon modifiable risk factors, such as the nutritional status, and potentially lower the risk of postoperative complications. However, the literature on perioperative optimization in HF comes mainly from anesthesiology and focuses on intra- and immediate postoperative management, when it may be too late to intervene and alter the outcome. Interestingly, guidelines on the nutritional evaluation and management of patients prior to non-cardiac surgery are available, but very limited literature is published concerning cardiac surgery, and no data exists with respect to LVAD surgery. The investigators plan to evaluation of the impact of preoperative nutrition intervention.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* hospitalized
* undergoing LVAD therapy (enrolled at time of acceptance)

Exclusion Criteria:

* intubated
* congenital heart disease
* infiltrative cardiomyopathy
* unable to tolerate oral nutrition
* surgery expected in <5 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Alpha Diversity (Baseline and Day 5) | Baseline and Day 5
  Change in alpha diversity (a measure of microbiome diversity applicable to a single sample) in collected stool samples.
Change in Alpha Diversity (Baseline and Pre-VAD) | Baseline and Pre-VAD (approximately Day 0-5)
  Change in alpha diversity (a measure of microbiome diversity applicable to a single sample) in collected stool samples.
Change in Alpha Diversity (Baseline and Discharge) | Baseline and Discharge (approximately Day 25)
  Change in alpha diversity (a measure of microbiome diversity applicable to a single sample) in collected stool samples.
Change in Alpha Diversity (Baseline and Post-Discharge Follow-up) | Baseline and Post-Discharge Follow-up (approximately Day 55)
  Change in alpha diversity (a measure of microbiome diversity applicable to a single sample) in collected stool samples.
Change in Microbial Gene Count (Baseline and Day 5) | Baseline and Day 5
  Change in microbial gene count as measured in stool samples.
Change in Microbial Gene Count (Baseline and Pre-VAD) | Baseline and Pre-VAD (approximately Day 0-5)
  Change in microbial gene count as measured in stool samples.
Change in Microbial Gene Count (Baseline and Discharge) | Baseline and Discharge (approximately Day 25)
  Change in microbial gene count as measured in stool samples.
Change in Microbial Gene Count (Baseline and Post-Discharge Follow-up) | Baseline and Post-Discharge Follow-up (approximately Day 55)
  Change in microbial gene count as measured in stool samples.
Change in C-Reactive Protein (CRP) (Baseline and Day 5) | Baseline and Day 5
  Change in biomarker CRP as measured in blood samples.
Change in C-Reactive Protein (CRP) (Baseline and Pre-VAD) | Baseline and Pre-VAD (approximately Day 0-5)
  Change in biomarker CRP as measured in blood samples.
Change in C-Reactive Protein (CRP) (Baseline and Discharge) | Baseline and Discharge (approximately Day 25)
  Change in biomarker CRP as measured in blood samples.
Change in C-Reactive Protein (CRP) (Baseline and Post-Discharge Follow-up) | Baseline and Post-Discharge Follow-up (approximately Day 55)
  Change in biomarker CRP as measured in blood samples.
Change in N-terminal (NT)-pro hormone BNP (NT-proBNP) (Baseline and Day 5) | Baseline and Day 5
  Change in biomarker NT-proBNP as measured in blood samples.
Change in N-terminal (NT)-pro hormone BNP (NT-proBNP) (Baseline and Pre-VAD) | Baseline and Pre-VAD (approximately Day 0-5)
  Change in biomarker NT-proBNP as measured in blood samples.
Change in N-terminal (NT)-pro hormone BNP (NT-proBNP) (Baseline and Discharge) | Baseline and Discharge (approximately Day 25)
  Change in biomarker NT-proBNP as measured in blood samples.
Change in N-terminal (NT)-pro hormone BNP (NT-proBNP) (Baseline and Post-Discharge Follow-up) | Baseline and Post-Discharge Follow-up (approximately Day 55)
  Change in biomarker NT-proBNP as measured in blood samples.
Change in lipopolysaccharide (LPS) (Baseline and Day 5) | Baseline and Day 5
  Change in biomarker LPS as measured in blood samples.
Change in lipopolysaccharide (LPS) (Baseline and Pre-VAD) | Baseline and Pre-VAD (approximately Day 0-5)
  Change in biomarker LPS as measured in blood samples.
Change in lipopolysaccharide (LPS) (Baseline and Discharge) | Baseline and Discharge (approximately Day 25)
  Change in biomarker LPS as measured in blood samples.
Change in lipopolysaccharide (LPS) (Baseline and Post-Discharge Follow-up) | Baseline and Post-Discharge Follow-up (approximately Day 55)
  Change in biomarker LPS as measured in blood samples.
Change in Tumor Necrosis Factor (TNF) (Baseline and Day 5) | Baseline and Day 5
  Change in biomarker TNF as measured in blood samples.
Change in Tumor Necrosis Factor (TNF) (Baseline and Pre-VAD) | Baseline and Pre-VAD (approximately Day 0-5)
  Change in biomarker TNF as measured in blood samples.
Change in Tumor Necrosis Factor (TNF) (Baseline and Discharge) | Baseline and Discharge (approximately Day 25)
  Change in biomarker TNF as measured in blood samples.
Change in Tumor Necrosis Factor (TNF) (Baseline and Post-Discharge Follow-up) | Baseline and Post-Discharge Follow-up (approximately Day 55)
  Change in biomarker TNF as measured in blood samples.
Change in Interleukin 6 (IL-6) (Baseline and Day 5) | Baseline and Day 5
  Change in biomarker IL-6 as measured in blood samples.
Change in Interleukin 6 (IL-6) (Baseline and Pre-VAD) | Baseline and Pre-VAD (approximately Day 0-5)
  Change in biomarker IL-6 as measured in blood samples.
Change in Interleukin 6 (IL-6) (Baseline and Discharge) | Baseline and Discharge (approximately Day 25)
  Change in biomarker IL-6 as measured in blood samples.
Change in Interleukin 6 (IL-6) (Baseline and Post-Discharge Follow-up) | Baseline and Post-Discharge Follow-up (approximately Day 55)
  Change in biomarker IL-6 as measured in blood samples.
Change in Interleukin 10 (IL-10) (Baseline and Day 5) | Baseline and Day 5
  Change in biomarker IL-10 as measured in blood samples.
Change in Interleukin 10 (IL-10) (Baseline and Pre-VAD) | Baseline and Pre-VAD (approximately Day 0-5)
  Change in biomarker IL-10 as measured in blood samples.
Change in Interleukin 10 (IL-10) (Baseline and Discharge) | Baseline and Discharge (approximately Day 25)
  Change in biomarker IL-10 as measured in blood samples.
Change in Interleukin 10 (IL-10) (Baseline and Post-Discharge Follow-up) | Baseline and Post-Discharge Follow-up (approximately Day 55)
  Change in biomarker IL-10 as measured in blood samples.
Change in Short-Chain Fatty Acids (Baseline and Day 5) | Baseline and Day 5
  Change in short-chain fatty acids as measured in blood samples.
Change in Short-Chain Fatty Acids (Baseline and Pre-VAD) | Baseline and Pre-VAD (approximately Day 0-5)
  Change in short-chain fatty acids as measured in blood samples.
Change in Short-Chain Fatty Acids (Baseline and Discharge) | Baseline and Discharge (approximately Day 25)
  Change in short-chain fatty acids as measured in blood samples.
Change in Short-Chain Fatty Acids (Baseline and Post-Discharge Follow-up) | Baseline and Post-Discharge Follow-up (approximately Day 55)
  Change in short-chain fatty acids as measured in blood samples.

SECONDARY OUTCOMES:
Post-LVAD Infections | Day 25
  Number and type of infections experienced during index hospitalization following LVAD implantation
Post-LVAD Length of Stay in intensive care unit | Day 25
  Number of days spent in intensive care unit following LVAD implantation.
Post-LVAD Mortality | Up to 2 years
  Number of participant deaths.

CONTACTS AND LOCATIONS:
Overall Officials: Melana Yuzefpolskaya, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savarese G, Lund LH. Global Public Health Burden of Heart Failure. Card Fail Rev. 2017 Apr;3(1):7-11. doi: 10.15420/cfr.2016:25:2. PMID 28785469
- [Background] Roger VL. Epidemiology of heart failure. Circ Res. 2013 Aug 30;113(6):646-59. doi: 10.1161/CIRCRESAHA.113.300268. PMID 23989710
- [Background] Francis GS, Benedict C, Johnstone DE, Kirlin PC, Nicklas J, Liang CS, Kubo SH, Rudin-Toretsky E, Yusuf S. Comparison of neuroendocrine activation in patients with left ventricular dysfunction with and without congestive heart failure. A substudy of the Studies of Left Ventricular Dysfunction (SOLVD). Circulation. 1990 Nov;82(5):1724-9. doi: 10.1161/01.cir.82.5.1724. PMID 2146040
- [Background] Munger MA, Johnson B, Amber IJ, Callahan KS, Gilbert EM. Circulating concentrations of proinflammatory cytokines in mild or moderate heart failure secondary to ischemic or idiopathic dilated cardiomyopathy. Am J Cardiol. 1996 Apr 1;77(9):723-7. doi: 10.1016/s0002-9149(97)89206-5. PMID 8651123
- [Background] Testa M, Yeh M, Lee P, Fanelli R, Loperfido F, Berman JW, LeJemtel TH. Circulating levels of cytokines and their endogenous modulators in patients with mild to severe congestive heart failure due to coronary artery disease or hypertension. J Am Coll Cardiol. 1996 Oct;28(4):964-71. doi: 10.1016/s0735-1097(96)00268-9. PMID 8837575
- [Background] Luedde M, Winkler T, Heinsen FA, Ruhlemann MC, Spehlmann ME, Bajrovic A, Lieb W, Franke A, Ott SJ, Frey N. Heart failure is associated with depletion of core intestinal microbiota. ESC Heart Fail. 2017 Aug;4(3):282-290. doi: 10.1002/ehf2.12155. Epub 2017 Apr 21. PMID 28772054
- [Background] Kummen M, Mayerhofer CCK, Vestad B, Broch K, Awoyemi A, Storm-Larsen C, Ueland T, Yndestad A, Hov JR, Troseid M. Gut Microbiota Signature in Heart Failure Defined From Profiling of 2 Independent Cohorts. J Am Coll Cardiol. 2018 Mar 13;71(10):1184-1186. doi: 10.1016/j.jacc.2017.12.057. No abstract available. PMID 29519360
- [Background] Sandek A, Bauditz J, Swidsinski A, Buhner S, Weber-Eibel J, von Haehling S, Schroedl W, Karhausen T, Doehner W, Rauchhaus M, Poole-Wilson P, Volk HD, Lochs H, Anker SD. Altered intestinal function in patients with chronic heart failure. J Am Coll Cardiol. 2007 Oct 16;50(16):1561-9. doi: 10.1016/j.jacc.2007.07.016. Epub 2007 Oct 1. PMID 17936155
- [Background] Schorghuber M, Fruhwald S. Effects of enteral nutrition on gastrointestinal function in patients who are critically ill. Lancet Gastroenterol Hepatol. 2018 Apr;3(4):281-287. doi: 10.1016/S2468-1253(18)30036-0. Epub 2018 Mar 7. PMID 29533200
- [Background] Lin H, Zhang H, Lin Z, Li X, Kong X, Sun G. Review of nutritional screening and assessment tools and clinical outcomes in heart failure. Heart Fail Rev. 2016 Sep;21(5):549-65. doi: 10.1007/s10741-016-9540-0. PMID 26920682
- [Background] Al-Najjar Y, Clark AL. Predicting outcome in patients with left ventricular systolic chronic heart failure using a nutritional risk index. Am J Cardiol. 2012 May 1;109(9):1315-20. doi: 10.1016/j.amjcard.2011.12.026. Epub 2012 Feb 13. PMID 22335857
- [Background] Sze S, Zhang J, Pellicori P, Morgan D, Hoye A, Clark AL. Prognostic value of simple frailty and malnutrition screening tools in patients with acute heart failure due to left ventricular systolic dysfunction. Clin Res Cardiol. 2017 Jul;106(7):533-541. doi: 10.1007/s00392-017-1082-5. Epub 2017 Feb 15. PMID 28204965
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, MacFie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery Society. Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):783-800. doi: 10.1016/j.clnu.2012.08.013. Epub 2012 Sep 28. PMID 23099039
- [Background] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Background] Yuzefpolskaya M, Bohn B, Nasiri M, Zuver AM, Onat DD, Royzman EA, Nwokocha J, Mabasa M, Pinsino A, Brunjes D, Gaudig A, Clemons A, Trinh P, Stump S, Giddins MJ, Topkara VK, Garan AR, Takeda K, Takayama H, Naka Y, Farr MA, Nandakumar R, Uhlemann AC, Colombo PC, Demmer RT. Gut microbiota, endotoxemia, inflammation, and oxidative stress in patients with heart failure, left ventricular assist device, and transplant. J Heart Lung Transplant. 2020 Sep;39(9):880-890. doi: 10.1016/j.healun.2020.02.004. Epub 2020 Feb 13. PMID 32139154